CLINICAL TRIAL: NCT00444899
Title: Clinical and Economic Benefits of Cardiovascular Risk Management by a Dietician in Diabetic Patients
Brief Title: Clinical and Economic Benefits of Cardiovascular Risk Management by a Dietician in Type 2 Diabetes Patients
Acronym: GRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocrinologist, researcher, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRA3840020
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Intensive treatment; dietician
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive treatment (Experimental): Submitted to an intensive follow-up by the dietician.
  Interventions: Behavioral: Intensive treatment
- Usual treatment (Active Comparator): Subjects will remain under the care of their endocrinologist and/or general practitioner.
  Interventions: Other: Normal follow-up

INTERVENTIONS:
Behavioral: Intensive treatment — Subjects will be followed by the dietician in combination with his/her endocrinologist. Diet, physical activity, smoking cessation and drug prescriptions will be used to treat subjects.
  Arms: Intensive treatment
Other: Normal follow-up — Subject will continue to be followed by their endocrinologist and general practitioner as they already do.
  Arms: Usual treatment

SUMMARY:
Worldwide, health systems and practitioners are facing obesity epidemics. High blood pressure, dyslipidemia and diabetes prevalence will explode during the 21st century.

The two main objectives of this 2-year controlled prospective study are:

1. to demonstrate that, for patients with high blood pressure, diabetes and dyslipidemia, dietician conducted survey and management in combination with annual endocrinologist follow-up enable both attainment and maintenance of recommended blood pressure, glycemic and lipid goals, as well as smoking cessation;
2. to demonstrate that dietician management is more cost effective than conventional care provided by general practitioners and endocrinologists.

Results are expected to show significantly different cardiovascular risk profiles (BMI and waist circumference, systolic and diastolic blood pressure, LDL-C, triglycerides and Total cholesterol/HDL ratio, HbA1c, smoking) between baseline and after 2 years follow-up. Sample size was determined in order to show statistically significant differences between the two groups.

Results will document for the benefit of care givers, health economists and policy makers alike an innovative and integrated model of care which is expected to be effective at the patient level as well as cost effective with respect to the increasing financial burden of diabetes on the health system.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > 7%
* More than 2 follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Lipid profile | 36 months
Blood pressure | 36 months
HbA1c | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Perron, MD, MSc, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche clinique Étienne-Le Bel du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No